CLINICAL TRIAL: NCT04883333
Title: A Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of LEO 153339 in Healthy Subjects
Brief Title: A Single and Multiple Ascending-dose Trial of LEO 153339 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0200-1495; 2020-005748-51 (EudraCT Number); U1111-1283-2001 (Other: World Health Organization (WHO))
Record Dates: First submitted 2021-05-11; First posted 2021-05-12 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Cohort A1 LEO 153339 (Experimental): Single ascending dose (Part 1)
  Interventions: Drug: LEO 153339
- Cohort A2 LEO 153339 (Experimental): Single ascending dose (Part 1)
  Interventions: Drug: LEO 153339
- Cohort A3 LEO 153339 (Experimental): Single ascending dose (Part 1)
  Interventions: Drug: LEO 153339
- Cohort A4 LEO 153339 (Experimental): Single ascending dose (Part 1)
  Interventions: Drug: LEO 153339
- Cohort A5 LEO 153339 (Experimental): Single ascending dose (Part 1)
  Interventions: Drug: LEO 153339
- Cohort A6 LEO 153339 (Experimental): Single ascending dose (Part 1)
  Interventions: Drug: LEO 153339
- Cohort A7 LEO 153339 (Experimental): Single ascending dose (Part 1)
  Interventions: Drug: LEO 153339
- Cohort B1 LEO 153339 (Experimental): Single ascending dose (Part 1)
  Interventions: Drug: LEO 153339
- All SAD cohorts placebo (Placebo Comparator): Single ascending dose (Part 1), all participants receiving placebo in Cohorts A1-A7 and B1
  Interventions: Drug: Placebo
- Cohort C1 LEO 153339 (Experimental): Multiple ascending doses (Part 2)
  Interventions: Drug: LEO 153339
- Cohort C2 LEO 153339 (Experimental): Multiple ascending doses (Part 2)
  Interventions: Drug: LEO 153339
- Cohort C3 LEO 153339 (Experimental): Multiple ascending doses (Part 2)
  Interventions: Drug: LEO 153339
- Cohort C4 LEO 153339 (Experimental): Multiple ascending doses (Part 2)
  Interventions: Drug: LEO 153339
- Cohort C5 LEO 153339 (Experimental): Multiple ascending doses (Part 2)
  Interventions: Drug: LEO 153339
- Cohort C6 LEO 153339 (Experimental): Multiple ascending doses (Part 2)
  Interventions: Drug: LEO 153339
- All MAD cohorts placebo (Placebo Comparator): Multiple ascending doses (Part 2, all participants receiving placebo in Cohorts C1-C6)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LEO 153339 — LEO 153339
  Arms: Cohort A1 LEO 153339; Cohort A2 LEO 153339; Cohort A3 LEO 153339; Cohort A4 LEO 153339; Cohort A5 LEO 153339; Cohort A6 LEO 153339; Cohort A7 LEO 153339; Cohort B1 LEO 153339; Cohort C1 LEO 153339; Cohort C2 LEO 153339; Cohort C3 LEO 153339; Cohort C4 LEO 153339; Cohort C5 LEO 153339; Cohort C6 LEO 153339
Drug: Placebo — Placebo
  Arms: All MAD cohorts placebo; All SAD cohorts placebo

SUMMARY:
This is a first-in-human study in adult healthy participants consisting of two parts. In Part 1, participants will receive one dose of study drug (LEO 153339) or placebo; in Part 2, participants will receive multiple doses of study drug or placebo.

The participants will stay in the clinic for 6 days (Part 1) or for 12 days (Part 2) to have the study doctor assess their safety and to investigate how quickly and to what extent LEO 153339 (and the breakdown product) is absorbed, transported, and eliminated from the body.

The purpose is to assess the safety and tolerability of LEO 153339 when compared to a placebo with no active ingredient.

ELIGIBILITY:
Main Inclusion Criteria:

* Healthy adult males and females.
* Age between 18 and 65 years (both inclusive) at screening.
* A body mass index (BMI) between 18.0 and 32.0 kg/m² (both inclusive).
* In good health at screening and/or check-in (Day -2 and Day -1) as judged by the investigator based on medical history, physical examination, vital signs, 12 lead electrocardiogram (ECG), and clinical laboratory evaluations.

Main Exclusion Criteria:

* Male participants sexually active with a woman of childbearing potential who are not willing to use a barrier method of contraception (e.g. condom) from the time of first dose of investigational medicinal product (IMP) until 3 months after the last dose, in conjunction with this female partner using a highly effective form of contraception. For vasectomised male participants, male participants with a female partner with bilateral tubal occlusion or ligation, and heterosexually abstinent male participants (when this is in line with the preferred and usual life style of the participant and not just being without a current partner), no additional contraception is required.
* Female participants who are pregnant, lactating, or of childbearing potential.
* Any surgical or medical condition or cholecystectomy which might significantly alter the absorption, distribution, metabolism, or excretion of any drug.
* Positive polymerase chain reaction (PCR) test for coronavirus disease 2019 (COVID-19) at Day -2 or Day -1 or within 8 weeks prior to screening or check-in, or contact with COVID-19 positive (or suspected) persons within 14 days prior to first dose.
* Treatment with any prescribed or non-prescribed systemic or topical medication within 7 days prior to the first dose of IMP (excluding paracetamol; including herbal remedies), unless, in the opinion of the investigator and the sponsor, the medication will not interfere with the trial procedures or compromise safety.
* Treatment with any non-marketed drug substance (that is, an agent which has not yet been made available for clinical use following registration) within 3 months prior to the first dose of IMP.
* ECG with QT interval corrected for heart rate using Fridericia's formula (QTcF) >450 msec confirmed by repeat measurement at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events per subject. | 4 days per subject (Part 1); 10 days per subject (Part 2)
  An adverse event will be considered treatment emergent if started after the first dose of investigational medicinal product (IMP) or if started before the first dose of IMP and worsened in severity after first dose of IMP.

SECONDARY OUTCOMES:
Plasma concentration of LEO 153339 and LEO 159074 obtained from 0 to 72 hours post-dose in subjects from the single ascending-dose (SAD) cohorts. | 72 hours per subject
  The pharmacokinetics of LEO 153339 and LEO 159074 will be evaluated in plasma.
Plasma concentration of LEO 153339 and LEO 159074 obtained from Day 1 to Day 7 post-dose with PK profiles on Day 1, Day 5, and Day 7 in subjects from the multiple ascending-dose (MAD) cohorts. | 10 days per subject
  The pharmacokinetics (PK) of LEO 153339 and LEO 159074 will be evaluated in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (1):
- LEO Pharma Investigational Site, Groningen, NZ, Netherlands

IPD SHARING:
Plan to Share IPD: No